CLINICAL TRIAL: NCT01224054
Title: Food Tolerance in Patients Submitted to Bariatric Surgery
Brief Title: Food and Gastrointestinal Habits After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Bruno Geloneze, University of Campinas, Brazil (UNICAMP)
Other Study IDs: LIMED0009; CEP 289/2008 (Other: Ethics Committee of Unicamp)
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Bariatric Surgeries
Keywords: Tolerance alimentary; Morbid obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bypass gastric: The mixed surgery which combine the gastric reduction with some degree of disabsorption
- Biliopancreatic diversion: The mal-absorptive surgery which reduce the intestinal absorption of food
- Duodenal exclusion: This surgery provides disabsortion by duodenal derivation maintaining an intact stomach

SUMMARY:
The worldwide epidemic of overweight and obesity affects about 1.7 billion people around the world. Since 1991, many international medical societies have established as recommendation for bariatric surgery the unsuccessful clinical treatment in patients with IMC > 40Kg/m2 or IMC > 35Kg/m2 in the cases with serious co-morbidities related to the possible reversion of them with the lose of weight due to the surgery. In front of the new anatomical condition from the gastrointestinal tract the patients present changes in food preferences and in the food intake, which include modifications in food choices, perception of hungry and satiety and in the tolerance to determinate food. These changes in food intake of the patients are observed mostly in the first year after the surgery an adaptive phase to a new condition.

DETAILED DESCRIPTION:
After the new anatomical condition of the gastrointestinal tract, provided by bariatric surgery leads patients to experience changes in food intake and behavior. The aim of this study was to assess alimentary habits, food intolerances and gastrointestinal symptoms in patients who underwent bariatric and metabolic procedures: Roux-en-Y gastric bypass, biliopancreatic diversion and duodenal exclusion. We studied 34 patients of both sexes, from outpatient clinics in Surgery of Obesity and the Metabolic Surgery at University of Campinas. They were submitted to bypass gastric in Roux-en-Y (n=15), biliopancreatic diversion (n=9) and duodenal exclusion (n=10). Validated questionnaire for assessment of food tolerance was applied in patients with more than six months of follow-up after surgery addressing diet and gastrointestinal symptoms. The descriptive and comparative analyses were performed by analysis of variance and bivariate correlation. In patients who underwent to bypass gastric food intolerance was greats regarding to ingestion of rice (33%) and red meat (33%) in comparison to others groups. The flatulence and diarrhea were more prevalent in patients who underwent biliopancreatic diversion. The vomiting was more prevalent in patients who underwent gastric bypass. Each procedure presents peculiarities to the anatomical and functional changes that affect the food absorption. This may have negative effects on the nutritional status of patients and affect the quality of life. The nutritional therapy for each individual procedure may assist in the management of clinical concerns of operated patients

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted of bypass gastric, biliopancreatic diversion and duodenal exclusion

Exclusion Criteria:

* Presenting no diseases that could compromise their nutritional status, such as liver disease, kidney or cancer.

Ages: 24 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: It was studied 34 patients (15 males, 19 female), ranging from 24 to 62 years old, who underwent bariatric surgery: gastric bypass (n=15), biliopancreatic diversion (n=9) or metabolic surgery: duodenal exclusion (n=10) with more than six months of follow-up postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Food tolerance in patients submitted to bariatric surgery | After 1 to 5 years of bariatric surgeries
  This study aims to assess habits and food intolerances and gastrointestinal symptoms in patients who underwent bariatric surgery: Roux-en-Y gastric bypass, biliopancreatic diversion and metabolic surgery: duodenal exclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Geloneze, Principal Investigator — University of Campinas (UNICAMP); Daniela Tezoto, Study Chair — +55-19-3521-8589; Éliton Chaim, Study Chair — University of Campinas (UNICAMP); Marcelo Lima, Study Chair — University of Campinas (UNICAMP); Sylka Geloneze, Study Chair — University of Campinas (UNICAMP); José Carlos Pareja, Study Chair — University of Campinas (UNICAMP); Vanessa Coutinho, Study Chair — Gama Filho University
Locations (1):
- LIMED - Laboratory of Investigation on Metabolism and Diabetes/Gastrocentro/University of Campinas (UNICAMP), Campinas, São Paulo, Brazil